CLINICAL TRIAL: NCT00399321
Title: A Pilot Study of Bone Mineral Density in Postmenopausal Women After Treatment for Breast Cancer
Status: Completed | Type: Observational
Sponsor: University of Michigan Rogel Cancer Center (Other)
Collaborators: Susan G. Komen Breast Cancer Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: UMCC 2006.016; HUM 3457
Record Dates: First submitted 2006-11-10; First posted 2006-11-14 (Estimated); Last update posted 2017-07-05 (Actual); Status verified 2017-07

CONDITIONS: Postmenopausal Bone Loss; Breast Cancer
Keywords: Post menopause women receiving adjuvant care
MeSH Terms: conditions — Osteoporosis, Postmenopausal; Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — refer to protocol
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The main purpose of this study is to see what levels of Bone Mineral Density post-menopausal women with breast cancer have, and to see if the level of Bone Mineral Density changes during a women's treatment after her surgery.

This trial studies changes in Bone Mineral Density and markers of of bone activity in post-menopausal women receiving treatment for early stage breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Documented diagnosis of breast cancer
* Last menstrual period occurring more than 5 years ago
* Non-metastatic breast cancer tumor with the diagnosis of Tis, Tl-T4, N0-3, M0
* DCIS is allowed, but LCIS (only) is not

Exclusion Criteria:

* Any metabolic bone disease other than postmenopausal osteoporosis or osteopenia
* Use of systemic gonadal hormonal medications or supplements within the past 24 months
* Prior use of tamoxifen or raloxifene is permitted if the medication was discontinued more than 24 months prior to the diagnosis of breast cancer.
* No adjuvant antiestrogen, antineoplastic, therapies are permitted on study.
* Chronic use of systemic steroids for disease process other than breast cancer chemotherapy premedication or antiemetics
* History of rheumatoid arthritis, ankylosing spondylitis, hyperparathyroidism, renal osteodystrophy, moderate to severe inflammatory or autoimmune disease or newly diagnosed thyroid condition requiring titration of medications.
* Lobular carcinoma in situ or Stage IV breast cancer and patients with a concurrently active second malignancy other then adequately treated non-melanoma skin cancers or in situ cervical cancer.
* participation in other clinical trials that are measuring BMD as a study parameter
* Patients with conditions that are expected to distort BMD reading and make DEXA results unreliable
* Patients with concurrent medical or psychiatric conditions that would keep them from understanding and complying with this clinical trial.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women with breast cancer
Sampling Method: Non-Probability Sample
Enrollment: 9 (Actual)
Dates: Start 2006-04; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Changes in bone mineral density in post-menopausal women receiving treatment for early stage breast cancer. | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Cathy Van Poznak, MD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan, United States